CLINICAL TRIAL: NCT03417102
Title: ATLAS-INH: A Phase 3 Study to Evaluate the Efficacy and Safety of Fitusiran in Patients With Hemophilia A or B, With Inhibitory Antibodies to Factor VIII or IX
Brief Title: A Study of Fitusiran (ALN-AT3SC) in Severe Hemophilia A and B Patients With Inhibitors
Acronym: ATLAS-INH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC14768; 2016-001463-36 (EudraCT Number); ALN-AT3SC-003 (Other: Alnylam)
Record Dates: First submitted 2018-01-25; First posted 2018-01-31 (Actual); Results first posted 2021-12-21 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: RNAi therapeutic; Hemophilia A; Hemophilia B; Hemophilia A, Severe; Hemophilia B, Severe; Blood Coagulation Disorders, Inherited; Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; Factor VIII; Factor IX; Inhibitor; Bypassing agents; Coagulants; Fitusiran
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Blood Coagulation Disorders, Inherited; Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn; Genetic Diseases, X-Linked | interventions — fitusiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bypassing Agents (BPA) On-demand (Active Comparator): Participants received On-demand BPAs (use of these agents, as needed, for episodic bleeding episodes, and not on a regular regimen intended to prevent spontaneous bleeding) per Investigator discretion from Day 1 for treatment of breakthrough bleeding episodes, up to a total of 9 months.
  Interventions: Drug: Bypassing agents
- Fitusiran 80 mg Prophylaxis (Experimental): Participants received Fitusiran 80 mg subcutaneously (SC) as prophylaxis once monthly from Day 1, along with the on-demand BPAs (per investigator's discretion and within bleeding dosing guidelines) for treatment of breakthrough bleeding episodes, up to a total of 9 months.
  Interventions: Drug: fitusiran

INTERVENTIONS:
Drug: fitusiran — solution for injection; by subcutaneous (SC) injection
  Arms: Fitusiran 80 mg Prophylaxis
Drug: Bypassing agents — solution for injection; by intravenous (IV) injection
  Arms: Bypassing Agents (BPA) On-demand

SUMMARY:
The purpose of this study was to determine the frequency of bleeding episodes in participants receiving fitusiran as prophylactic treatment of hemophilia compared to participants who were assigned to continue with their regular medication. In addition, the study assessed safety, quality of life, pharmacodynamics (PD), and pharmacokinetics (PK).

DETAILED DESCRIPTION:
The duration of treatment with fitusiran was 9 months. The estimated total time on study, inclusive of screening, for each participant was up to 11 months for all participants who enroll in the extension study and participants in the on-demand arm who did not enroll in the extension study. The estimated total time on study was up to 17 months in fitusiran treatment arm participants who did not enroll in the extension study due to the requirement for up to an additional 6 months of follow-up monitoring for antithrombin levels.

ELIGIBILITY:
Inclusion Criteria:

* Males, greater than or equal to (>=) 12 years of age.
* Severe hemophilia A or B with inhibitors.

  * (Severity confirmed by a central laboratory where coagulation factor VIII (FVIII) level was less than (<)1% or factor IX (FIX) level was less than or equal to [<=]2% at Screening; Inhibitors defined as inhibitor titer of >=0.6 Bethesda units per milliliter [BU/mL] or as evidenced by medical records).
* A minimum of 6 bleeding episodes requiring BPA treatment within the last 6 months prior to screening.
* Willing and able to comply with the study requirements and to provide written informed consent and assent.

Exclusion Criteria:

* Known co-existing bleeding disorders other than hemophilia A or B.
* Antithrombin (AT) activity <60% at Screening.
* Co-existing thrombophilic disorder.
* Clinically significant liver disease.
* Active hepatitis C virus infection.
* HIV positive with a cluster of differentiation-4 count of <200 cells/microliter.
* History of arterial or venous thromboembolism.
* Inadequate renal function.
* History of multiple drug allergies or history of allergic reaction to an oligonucleotide or N-Acetylgalactosamine.
* History of intolerance to SC injection(s).
* Any other conditions or comorbidities that would make the participant unsuitable for enrollment or could interfere with participation in or completion of the study, per Investigator judgement.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2021-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, MD, Study Director — Sanofi
Locations (58):
- United States (12):
  - Investigational Site Number 0117, Phoenix, Arizona
  - Investigational Site Number 0139, Los Angeles, California
  - Investigational Site Number 0135, Orange, California
  - Investigational Site Number 0137, San Diego, California
  - Investigational Site Number 0128, Gainesville, Florida
  - Investigational Site Number 0115, Jacksonville, Florida
  - Investigational Site Number 0105, Miami, Florida
  - Investigational Site Number 0103, Tampa, Florida
  - Investigational Site Number 0119, New Orleans, Louisiana
  - Investigational Site Number 0136, Baltimore, Maryland
  - Investigational Site Number 0111, Las Vegas, Nevada
  - Investigational Site Number 0104, Philadelphia, Pennsylvania
- Australia (2):
  - Investigational Site Number 6101, Camperdown
  - Investigational Site Number 6104, Clayton
- Investigational Site Number 1102, Montreal, Canada
- China (5):
  - Investigational Site Number 8604, Beijing
  - Investigational Site Number 8602, Guangzhou
  - Investigational Site Number 8605, Hangzhou
  - Investigational Site Number 8603, Shanghai
  - Investigational Site Number 8601, Tianjin
- France (2):
  - Investigational Site Number 3303, Lyon
  - Investigational Site Number 3301, Rouen
- Germany (2):
  - Investigational Site Number 4905, Frankfurt am Main
  - Investigational Site Number 4906, Leipzig
- India (7):
  - Investigational Site Number 9102, Bangalore
  - Investigational Site Number 9108, India
  - Investigational Site Number 9104, Jaipur
  - Investigational Site Number 9106, Lucknow
  - Investigational Site Number 9103, Pune
  - Investigational Site Number 9111, Pune
  - Investigational Site Number 9105, Vellore
- Italy (2):
  - Investigational Site Number 3901, Florence
  - Investigational Site Number 3904, Padua
- Japan (2):
  - Investigational Site Number 8110, Japan
  - Investigational Site Number 8103, Kita Kyushu-Shi
- Malaysia (2):
  - Investigational Site Number 6003, Kota Kinabalu
  - Investigational Site Number 6004, Malaysia
- South Africa (3):
  - Investigational Site Number 2701, Parktown
  - Investigational Site Number 2703, Polokwane
  - Investigational Site Number 2702, Port Elizabeth
- South Korea (3):
  - Investigational Site Number 8202, Daejeon
  - Investigational Site Number 8203, Seoul
  - Investigational Site Number 8204, Seoul
- Investigational Site Number 3402, Madrid, Spain
- Taiwan (4):
  - Investigational Site Number 8803, Changhua
  - Investigational Site Number 8804, Dawan
  - Investigational Site Number 8805, Dawan
  - Investigational Site Number 8801, Taipei
- Turkey (Türkiye) (6):
  - Investigational Site Number 9002, Adana
  - Investigational Site Number 9004, Akdeniz
  - Investigational Site Number 9001, Ankara
  - Investigational Site Number 9005, Istanbul
  - Investigational Site Number 9003, Izmir
  - Investigational Site Number 9006, Turkey
- Ukraine (3):
  - Investigational Site Number 8003, Kyiv
  - Investigational Site Number 8001, Kyiv
  - Investigational Site Number 8002, Lviv
- Investigational Site Number 4407, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Young G, Srivastava A, Kavakli K, Ross C, Sathar J, You CW, Tran H, Sun J, Wu R, Poloskey S, Qiu Z, Kichou S, Andersson S, Mei B, Rangarajan S. Efficacy and safety of fitusiran prophylaxis in people with haemophilia A or haemophilia B with inhibitors (ATLAS-INH): a multicentre, open-label, randomised phase 3 trial. Lancet. 2023 Apr 29;401(10386):1427-1437. doi: 10.1016/S0140-6736(23)00284-2. Epub 2023 Mar 29. PMID 37003287
- [Derived] The Lancet Haematology. The role of conferences in tackling inequalities. Lancet Haematol. 2022 Feb;9(2):e81. doi: 10.1016/S2352-3026(22)00008-4. No abstract available. PMID 35114155
- [Derived] Del Pozo Martin Y. 2021 ASH annual meeting. Lancet Haematol. 2022 Feb;9(2):e92-e93. doi: 10.1016/S2352-3026(21)00384-7. Epub 2021 Dec 16. No abstract available. PMID 34922648

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 58 centers in 17 countries. A total of 85 participants were screened between 14 February 2018 to 19-Mar-2021, of which 25 participants were screen failure. Screen failures were mainly due to the presence of clinically significant liver disease. A total of 60 participants were enrolled in the study.
Pre-assignment Details: 57 participants randomized in 2:1 ratio to fitusiran prophylaxis and on-demand arms; stratified by number of bleeding episodes prior to Screening (<=10 vs >10). 3 participants from China were treated with fitusiran but not randomized. These participants were considered in fitusiran prophylaxis arm for safety analysis, but not in any other analysis.
Period: Overall Study
Arm/Group | Bypassing Agents (BPA) On-demand | Fitusiran 80 mg Prophylaxis
Started | 19 | 38
Safety Analysis Set (Participants received at least 1 dose of study drug or randomized to on-demand arm, analyzed per treatment received.) | 19 | 41 (3 participants were non-randomized but treated with Fitusiran considered in this arm for safety.)
Completed | 19 | 33
Not Completed | 0 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Related to Coronavirus Pandemic (Covid-19) | 0 | 3
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent-to-Treat (ITT) population which included all randomized participants who were analyzed according to the randomized treatment arm.
Arm/Group | Bypassing Agents (BPA) On-demand | Fitusiran 80 mg Prophylaxis | Total Title
Number analyzed (Participants) | 19 | 38 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (13.1) | 26.8 (9.8) | 28.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 19 | 38 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 26 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 10 | 16
  Other | 0 | 1 | 1
  Multiple | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Estimated Annualized Bleeding Rate (ABR) for Treated Bleeds During the Efficacy Period
Description: ABR for a participant during efficacy period (EP) was defined as annualized number of bleeding episodes during EP annualized to a 1-year interval of time. Treated Bleeding episode: any occurrence of hemorrhage that required administration of BPA or factor. It started from first sign of a bleed and ended no more than 72 hours after last treatment for bleed, within which any symptoms of bleeding at same location or injections less than or equal to 72 hours apart were considered the same bleeding episode. EP was defined as time duration starting from Day 29 when antithrombin (AT) lowering capacity of fitusiran had achieved therapeutic target range to the earliest of (Day 246 or last day of bleeding follow up) (maximum duration of EP: from Day 29 to Day 246). This outcome measure (OM) represents estimated results (i.e., results received by applying negative binomial [NB] regression model on data collected during EP).
Time Frame: From Day 29 up to Day 246 or up to the last day of bleeding follow up (any day up to Day 246), whichever was the earliest
Population: Analysis was performed on ITT population.
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Bypassing Agents (BPA) On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 19 | 38
episodes per participant per year | 18.071 [10.598 to 30.812] | 1.666 [1.014 to 2.736]
Statistical Analysis 1: Comparison: Bypassing Agents (BPA) On-demand vs Fitusiran 80 mg Prophylaxis; Test type: Superiority; p < 0.0001, Negative binomial regression model — P-value derived from NB regression model, accounted for different follow-up times during EP, with treatment arm and randomization strata of number of bleeds in 6 months prior to study (<=10,>10) as fixed effects. Significance threshold was 0.05; ABR ratio = 0.092, 95% CI 2-sided [0.044 to 0.192]

2. Primary Outcome: Observed Annualized Bleeding Rate (ABR) for Treated Bleeds During the Efficacy Period
Description: ABR for a participant during EP was defined as annualized number of bleeding episodes during EP annualized to a 1-year interval of time. ABR= number of bleeding episodes during EP divided by total number of days during EP*365.25. A bleeding episode was defined as any occurrence of hemorrhage that required administration of BPA or factor. It started from the first sign of a bleed and ended no more than 72 hours after the last treatment for the bleed, within which any symptoms of bleeding at the same location or injections less than or equal to 72 hours apart were considered the same bleeding episode. EP was defined as time duration starting from Day 29 when the AT lowering capacity of fitusiran had achieved therapeutic target range to the earliest of (Day 246 or the last day of bleeding follow up) (maximum duration of EP: from Day 29 to Day 246). This OM represents observed results (i.e., descriptive statistics values based on the data which was collected during EP).
Time Frame: as for outcome 1
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | Bypassing Agents (BPA) On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 19 | 38
episodes per participant per year | 18.1 (14.9) | 1.7 (3.8)

3. Secondary Outcome: Estimated Annualized Bleeding Rate (ABR) for Treated Bleeds During the Treatment Period
Description: ABR for a participant during treatment period (TP) was defined as annualized number of bleeding episodes during TP annualized to a 1-year interval of time. Bleeding episode: any occurrence of hemorrhage that required administration of BPA or factor. It started from first sign of a bleed and ended no more than 72 hours after last treatment for bleed, within which any symptoms of bleeding at same location or injections less than or equal to 72 hours apart were considered the same bleeding episode. TP was sum of onset period (first 28 days after first dose of fitusiran) and EP (starting on Day 29 when AT lowering capacity of fitusiran had achieved therapeutic target range to earliest of [Day 246 or last day of bleeding follow up])(maximum duration of TP: from Day 1 to Day 246). This OM represents estimated results (i.e., results received by applying NB regression model on data collected during TP).
Time Frame: From Day 1 up to Day 246 or up to the last day of bleeding follow up (any day up to Day 246), whichever was the earliest
Population: Analysis was performed on ITT population.
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Bypassing Agents (BPA) On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 19 | 38
episodes per participant per year | 18.819 [11.541 to 30.687] | 2.024 [1.306 to 3.138]
Statistical Analysis 1: Comparison: Bypassing Agents (BPA) On-demand vs Fitusiran 80 mg Prophylaxis; Test type: Superiority; p < 0.0001, Negative binomial regression model — P-value derived from NB regression model, accounted for different follow-up times during TP, with treatment arm and randomization strata of number of bleeds in 6 months prior to study (<=10,>10) as fixed effects. Significance threshold was 0.05; ABR ratio = 0.108, 95% CI 2-sided [0.056 to 0.207]

4. Secondary Outcome: Observed Annualized Bleeding Rate (ABR) for Treated Bleeds During the Treatment Period
Description: ABR for a participant during TP was defined as annualized number of bleeding episodes during TP annualized to a 1-year interval of time. ABR= number of bleeding episodes during TP divided by total number of days during TP*365.25. Bleeding episode: any occurrence of hemorrhage that required administration of BPA or factor. It started from the first sign of a bleed and ended no more than 72 hours after last treatment for bleed, within which any symptoms of bleeding at the same location or injections less than or equal to 72 hours apart were considered the same bleeding episode. TP was sum of onset period (first 28 days after the first dose of fitusiran) and EP (starting on Day 29 when AT lowering capacity of fitusiran had achieved therapeutic target range to the earliest of [Day 246 or the last day of bleeding follow up]) (maximum duration of TP: from Day 1 to Day 246). This OM represents observed results (i.e., descriptive statistics values based on data collected during TP).
Time Frame: as for outcome 3
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | Bypassing Agents (BPA) On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 19 | 38
episodes per participant per year | 18.8 (15.4) | 2.0 (3.7)

5. Secondary Outcome: Estimated Annualized Spontaneous Bleeding Rate for Treated Bleeds During Efficacy Period
Description: Annualized spontaneous bleeding rate for a participant during EP was defined as annualized number of spontaneous bleeding episodes during EP annualized to a 1-year interval of time. Spontaneous bleeding episode was bleeding event that occurred for no apparent or known reason, particularly into joints, muscles, and soft tissues. It started from first sign of a bleed and ended no more than 72 hours after last treatment for the bleed, within which any symptoms of bleeding at the same location or injections less than or equal to 72 hours apart were considered the same bleeding episode. EP was defined as time duration starting from Day 29 when AT lowering capacity of fitusiran had achieved therapeutic target range to the earliest of (Day 246 or last day of bleeding follow up) (maximum duration of EP: from Day 29 to Day 246). This OM represents estimated results (i.e., results received by applying NB regression model on data collected during EP).
Time Frame: as for outcome 1
Population: Analysis was performed on ITT population.
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Bypassing Agents (BPA) On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 19 | 38
episodes per participant per year | 15.675 [9.281 to 26.471] | 0.872 [0.491 to 1.551]
Statistical Analysis 1: Comparison: Bypassing Agents (BPA) On-demand vs Fitusiran 80 mg Prophylaxis; Test type: Superiority; p < 0.0001, Negative binomial regression model — [p-value comment as in outcome 1, analysis 1]; ABR ratio = 0.056, 95% CI 2-sided [0.026 to 0.121]

6. Secondary Outcome: Observed Annualized Spontaneous Bleeding Rate for Treated Bleeds During the Efficacy Period
Description: ABR for participant during EP was defined as annualized number of spontaneous bleeding episodes during EP annualized to a 1-year interval of time. ABR=number of treated spontaneous bleeding episodes during EP divided by total number of days during EP*365.25. Spontaneous bleeding episode was bleeding event that occurred for no apparent or known reason, into joints, muscles, and soft tissues. It started from the first sign of a bleed and ended no more than 72 hours after the last treatment for bleed, within which any symptoms of bleeding at the same location or injections less than or equal to 72 hours apart were considered the same bleeding episode. EP: time duration starting from Day 29 when the AT lowering capacity of fitusiran had achieved therapeutic target range to earliest of (Day 246 or the last day of bleeding follow up) (maximum duration of EP: from Day 29 to Day 246). This OM represents observed results (i.e., descriptive statistics values based on data collected during EP).
Time Frame: as for outcome 1
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | Bypassing Agents (BPA) On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 19 | 38
episodes per participant per year | 15.6 (14.9) | 0.9 (2.0)

7. Secondary Outcome: Estimated Annualized Joint Bleeding Rate for Treated Bleeds During the Efficacy Period
Description: Annualized joint bleeding rate for a participant during EP was defined as annualized number of bleeding episodes during EP annualized to a 1-year interval of time. Joint bleeding episode was characterized by an unusual sensation in the joint ("aura") in combination with 1) increasing swelling or warmth over the skin, joint, 2) increased pain, or 3) progressive loss of range of motion or difficulty in using the limb as compared with Baseline. It started from first sign of a bleed and ended no more than 72 hours after last treatment for the bleed. EP was defined as time duration starting from Day 29 when the AT lowering capacity of fitusiran had achieved therapeutic target range to the earliest of (Day 246 or the last day of bleeding follow up) (maximum duration of EP: from Day 29 to Day 246). This OM presents estimated results (i.e., results received by applying NB regression model on data collected during EP).
Time Frame: as for outcome 1
Population: Analysis was performed on ITT population.
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Bypassing Agents (BPA) On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 19 | 38
episodes per participant per year | 13.759 [7.950 to 23.811] | 1.349 [0.798 to 2.280]
Statistical Analysis 1: Comparison: Bypassing Agents (BPA) On-demand vs Fitusiran 80 mg Prophylaxis; Test type: Superiority; p < 0.0001, Negative binomial regression model — [p-value comment as in outcome 1, analysis 1]; ABR ratio = 0.098, 95% CI 2-sided [0.046 to 0.210]

8. Secondary Outcome: Observed Annualized Joint Bleeding Rate for Treated Bleeds During the Efficacy Period
Description: Annualized joint bleeding rate for participant during EP was defined as annualized number of joint bleeding episodes during EP annualized to 1-year interval of time. ABR= number of treated joint bleeding episodes during EP divided by total number of days during EP*365.25. A joint bleeding episode was characterized by an unusual sensation in joint ("aura") in combination with 1) increasing swelling or warmth over skin, joint, 2) increased pain, or 3) progressive loss of range of motion or difficulty in using limb as compared with Baseline. It started from first sign of a bleed and ended no more than 72 hours after the last treatment for the bleed. EP: time duration starting from Day 29 when the AT lowering capacity of fitusiran had achieved therapeutic target range to the earliest of (Day 246 or last day of bleeding follow up) (maximum duration of EP: from Day 29 to Day 246). This OM presents observed results (i.e., descriptive statistics values based on data collected during EP).
Time Frame: as for outcome 1
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | Bypassing Agents (BPA) On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 19 | 38
episodes per participant per year | 13.8 (12.2) | 1.4 (3.4)

9. Secondary Outcome: Health-related Quality of Life (HRQOL): Change From Baseline in Haemophilia Quality of Life Questionnaire for Adults (Haem-A-QOL) Physical Health Domain Score at Month 9
Description: Haem-A-QoL: participant-reported questionnaire designed for adult participants (>=17 years of age) with hemophilia; and consisted of 46 items comprising 10 domains (physical health, feelings, view of yourself, sports and leisure, work and school, dealing with hemophilia, treatment, future, family planning, partnership and sexuality). Items were rated along five response options: never, rarely, sometimes, often, or all the time. Change from baseline in physical Health domain score was reported in this outcome measure. Raw score for physical health domain were transformed to a scale ranged from 0 to 100, where lower scores denoted better physical health.
Time Frame: Baseline (Day 1), Month 9
Population: Analysis was performed on ITT population. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Bypassing Agents (BPA) On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 17 | 32
score on a scale | -1.94 [-10.32 to 6.43] | -30.67 [-36.90 to -24.43]
Statistical Analysis 1: Comparison: Bypassing Agents (BPA) On-demand vs Fitusiran 80 mg Prophylaxis; Test type: Superiority; p < 0.0001, ANCOVA — Analysis of Covariance (ANCOVA) model included treatment arm and randomization strata of number of bleeds (<=10, > 10) as fixed effects, Baseline score as a covariate. Significance threshold was at 0.05; Least Square (LS) Mean difference = -28.72, 95% CI 2-sided [-39.07 to -18.37]

10. Secondary Outcome: Health-related Quality of Life (HRQOL): Change From Baseline in Haem-A-QOL Total Score at Month 9
Description: Haem-A-QoL: participant-reported questionnaire designed for adult participants (>=17 years of age) with hemophilia; and consisted of 46 items comprising 10 domains (physical health, feelings, view of yourself, sports and leisure, work and school, dealing with hemophilia, treatment, future, family planning, partnership and sexuality). Items were rated along five response options: never, rarely, sometimes, often, or all the time. Raw score for each domain were transformed to a scale ranged from 0 to 100, where lower scores denoted better health. Haem-A-QoL Total Score was average of all domain scores and ranged from 0 to 100, where lower scores denoted better quality of life.
Time Frame: Baseline (Day 1), Month 9
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Bypassing Agents (BPA) On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 17 | 31
score on a scale | -0.42 [-5.65 to 4.80] | -15.27 [-19.30 to -11.24]
Statistical Analysis 1: Comparison: Bypassing Agents (BPA) On-demand vs Fitusiran 80 mg Prophylaxis; Test type: Superiority; p < 0.0001, ANCOVA — ANCOVA model included treatment arm and randomization strata of number of bleeds (<=10, > 10) as fixed effects, Baseline score as a covariate. Significance threshold was at 0.05; LS Mean difference = -14.85, 95% CI 2-sided [-21.37 to -8.33]

11. Secondary Outcome: Estimated Annualized Bleeding Rate (ABR) for Treated Bleeds During the Onset Period
Description: ABR was annualized number of bleeding episodes during onset period per participant annualized to a 1-year interval of time. A treated bleeding episode was defined as any occurrence of hemorrhage that may required administration of BPA or factor. It started from the first sign of a bleed and ended no more than 72 hours after the last treatment for the bleed, within which any symptoms of bleeding at the same location or injections less than or equal to 72 hours apart were considered the same bleeding episode. The onset period was defined as time interval from Day 1 to the earlier of Day 28 or the last day of bleeding follow up. This OM represents estimated results (i.e., results received by applying NB regression model on data collected during onset period).
Time Frame: From Day 1 up to Day 28 or up to the last day of bleeding follow up (any day up to Day 28), whichever was the earliest
Population: Analysis was performed on ITT population.
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Bypassing Agents (BPA) On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 19 | 38
episodes per participant per year | 25.149 [15.819 to 39.981] | 4.426 [2.439 to 8.030]

12. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse Event (AE) was defined as any untoward medical occurrence in a participant who received study drug which did not necessarily have a causal relationship with the treatment. Treatment emergent AEs were defined as any AE with onset date after first dose of fitusiran in the fitusiran prophylaxis arm or after Day 1 visit in the BPA on-demand arm. A Serious AE (SAE) was defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability or incapacity, was a congenital anomaly or birth defect, or was a medically important event.
Time Frame: From Baseline (Day 1) up to 15 months (i.e. 9 months treatment period + 6-months follow-up)
Population: Analysis was performed on safety analysis set that included all participants who received at least 1 dose of study drug or were randomized to on-demand arm, analyzed according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Bypassing Agents (BPA) On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 19 | 41
Participants
  Any TEAE | 11 | 38
  Any TESAE | 5 | 7

ADVERSE EVENTS:
Time Frame: AE data were collected from Baseline (Day 1) up to 15 months (i.e., 9 months treatment period + 6-months follow-up).
Description: TEAEs: any AE with onset date after first dose of fitusiran in fitusiran prophylaxis arm or after Day 1 visit in the BPA on-demand arm. Analysis done on safety analysis set. Three participants who were treated with fitusiran but not randomized as per protocol addendum for China, were included in safety analysis for the fitusiran prophylaxis arm.
Arm/Group | Bypassing Agents (BPA) On-demand | Fitusiran 80 mg Prophylaxis
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/41
Serious Adverse Events (participants affected / at risk) | 5/19 | 7/41
Other Adverse Events (participants affected / at risk) | 8/19 | 32/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bypassing Agents (BPA) On-demand (N=19) | Fitusiran 80 mg Prophylaxis (N=41)
Tooth Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic Haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Spinal Vascular Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asymptomatic Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1)
Haematoma Infection (Infections and infestations) | 0 (0) | 1 (1)
Vascular Device Infection (Infections and infestations) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Subclavian Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Biliary Colic (Hepatobiliary disorders) | 0 (0) | 1 (2)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis Chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bypassing Agents (BPA) On-demand (N=19) | Fitusiran 80 mg Prophylaxis (N=41)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 13 (23)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 8 (16)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 5 (9)
Fibrin D Dimer Increased (Investigations) | 0 (0) | 3 (6)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 6 (9)
Prothrombin Fragment 1.2 Increased (Investigations) | 0 (0) | 3 (6)
Transaminases Increased (Investigations) | 0 (0) | 5 (6)
Headache (Nervous system disorders) | 1 (1) | 6 (9)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 6 (7)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (13)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Asymptomatic Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (5)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 6 (8)
Asthenia (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT03417102/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT03417102/SAP_001.pdf